CLINICAL TRIAL: NCT06862037
Title: Development of Elastic Net Regression-SMOTE Models to Predict Postoperative Gastroesophageal Reflux Symptom Resolution After Laparoscopic Nissen Fundoplication
Brief Title: Development of Machine Learning Models to Predict Postoperative GERD Symptom Resolution After Laparoscopic Nissen Fundoplication
Status: Active, not recruiting | Type: Observational
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Sungsoo Park, Professor, Korea University Anam Hospital
Other Study IDs: LNF-ML-D
Record Dates: First submitted 2025-03-02; First posted 2025-03-06 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-02

CONDITIONS: Gastroesophageal Reflux Disease (GERD); Gastroesophageal Reflux (GER)
Keywords: Gastroesophageal reflux disease; Laparoscopic Nissen fundoplication; Machine learning; Elastic Net regression; SMOTE; endoscopy; esophagogastroduodenoscopy; esophageal pH monitoring; manometry
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Symptom resolution group: Preoperative and postoperative gastroesophageal symptoms, including heartburn and regurgitation, were evaluated using the GERD-HRQL and the Korean version of the GERD questionnaire. Postoperative symptoms were assessed at 1, 3, 6, 9, and 12 months after laparoscopic Nissen fundoplication. Patients with more than a 70% improvement in symptoms at the last follow-up will be classified as the symptom resolution group.
  Interventions: Procedure: Laparoscopic Nissen fundoplication
- Symptom non-resolution group: Preoperative and postoperative gastroesophageal symptoms, including heartburn and regurgitation, were evaluated using the GERD-HRQL and the Korean version of the GERD questionnaire. Postoperative symptoms were assessed at 1, 3, 6, 9, and 12 months after laparoscopic Nissen fundoplication. Patients with less than a 70% improvement in symptoms at the last follow-up will be classified as the symptom non-resolution group.
  Interventions: Procedure: Laparoscopic Nissen fundoplication

INTERVENTIONS:
Procedure: Laparoscopic Nissen fundoplication — Laparoscopic Nissen fundoplication (LNF) is the most commonly performed anti-reflux surgery. LNF is performed in patients with GERD refractory to medication or those expected to require long-term medical treatment. During LNF, the fundus of the stomach is mobilized and wrapped 360 degrees around the lower esophagus to reinforce the lower esophageal sphincter (LES), preventing the reflux of gastric contents into the esophagus.

SUMMARY:
This study aims to develop machine learning models to predict postoperative gastroesophageal reflux symptom resolution after laparoscopic Nissen fundoplication using Elastic Net regression and synthetic minority oversampling technique (SMOTE).

DETAILED DESCRIPTION:
In patients with gastroesophageal reflux disease (GERD) refractory to medication or those expected to require long-term medical treatment, anti-reflux surgery (ARS), including Nissen fundoplication, has been performed. GERD is usually diagnosed as esophageal mucosal damage or pathological esophageal acid exposure. However, about 35% of patients with gastroesophageal reflux symptoms do not exhibit abnormal findings on esophagogastroduodenoscopy (EGD) and esophageal pH monitoring. Meanwhile, about 10% of patients with typical GERD symptoms and 30-50% of those with atypical GERD symptoms do not experience symptom improvement even after undergoing ARS. Therefore, the importance of predicting symptom improvement after ARS and appropriately selecting surgical candidates has been increasingly emphasized.

Though previous studies have suggested several predictors-including the length of the lower esophageal sphincter (LES), resting pressure of the LES, and bolus exposure time-to predict GERD symptom resolution after ARS, no model comprehensively integrated the results of EGD, esophageal pH monitoring, and manometry.

Elastic Net regression is a machine learning method that utilizes regularized regression analysis, combining L1 (Lasso) and L2 (Ridge) penalties. This approach makes the model relatively robust against overfitting and is suitable for datasets with a small sample size, a large number of variables, and severe multicollinearity. Synthetic minority oversampling technique (SMOTE) is a method that enhances the interpretability of the minority class in a model by oversampling minority class data using the k-nearest neighbors (k-NN) algorithm. Therefore, this study aims to develop machine learning models to predict postoperative gastroesophageal reflux symptom resolution after laparoscopic Nissen fundoplication using Elastic Net regression and SMOTE.

A total of 112 patients who underwent LNF between February 2017 to February 2023 will be included in this study. Preoperative and postoperative gastroesophageal symptoms, including heartburn and regurgitation, were evaluated using the GERD Health-Related Quality of Life (GERD-HRQL) questionnaire and the Korean version of the GERD questionnaire. Postoperative symptoms were assessed at 1, 3, 6, 9, and 12 months after surgery. Patients with more than a 70% improvement in symptoms at the last follow-up will be classified as the symptom resolution group. A total of 21 models will be developed to predict the resolution of heartburn, regurgitation, or atypical symptoms using the results of manometry, 24-hour esophageal pH monitoring, or both, with seven models for each symptom. All models will also incorporate the results of EGD. Elastic Net regression and the SMOTE method will be applied to oversample the minority class and develop the model. Model performance will be validated using 5-fold cross-validation. In addition to assessing model discrimination, calibration analysis will be performed to evaluate how well the predicted probabilities align with observed outcomes. The predictive performance of conventional predictors and possible predictors, including the length of LES, resting pressure of the LES, and bolus exposure time, will be compared with the model performance of the novel model.

ELIGIBILITY:
Inclusion Criteria:

1. patients with age greater than 19 years
2. patients who underwent laparoscopic Nissen fundoplication from February 2017 to February 2023
3. patients who answered the GERD-HRQL questionnaire or the Korean version of the GERD questionnaire to assess preoperative and postoperative gastroesophageal reflux symptoms
4. patients who underwent esophagogastroduodenoscopy before surgery
5. patients who underwent esophageal manometry, 24-hour esophageal pH monitoring, or both before surgery

Exclusion Criteria:

1. pregnant
2. patients who were lost to follow-up before 3 months after surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent laparoscopic Nissen fundoplication
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Model performance of novel models | Symptoms were assessed before surgery and at 1, 3, 6, 9, and 12 months after surgery
  A total of 21 models will be developed to predict the resolution of heartburn, regurgitation, or atypical symptoms using the results of manometry, 24-hour esophageal pH monitoring, or both, with seven models for each symptom. All models will also incorporate the results of EGD. Elastic Net regression and the SMOTE method will be applied to oversample the minority class and develop the model. Model performance including AUC, sensitivity (or recall), specificity, accuracy, precision, and F1 score will be validated using 5-fold cross-validation.

SECONDARY OUTCOMES:
Results from calibration analysis of novel models | Symptoms were assessed before surgery and at 1, 3, 6, 9, and 12 months after surgery
  A total of 21 models will be developed to predict the resolution of heartburn, regurgitation, or atypical symptoms using the results of manometry, 24-hour esophageal pH monitoring, or both, with seven models for each symptom. All models will also incorporate the results of EGD. Elastic Net regression and the SMOTE method will be applied to oversample the minority class and develop the model. Calibration analysis will be performed to evaluate how well the predicted probabilities align with observed outcomes.

OTHER OUTCOMES:
Predictive performance of conventional predictors and possible predictors | Symptoms were assessed before surgery and at 1, 3, 6, 9, and 12 months after surgery
  A total of 21 models will be developed to predict the resolution of heartburn, regurgitation, or atypical symptoms using the results of manometry, 24-hour esophageal pH monitoring, or both, with seven models for each symptom. All models will also incorporate the results of EGD. Elastic Net regression and the SMOTE method will be applied to oversample the minority class and develop the model. Model performance will be validated using 5-fold cross-validation. The predictive performance of conventional predictors and possible predictors, including the length of LES, resting pressure of the LES, and bolus exposure time, will be compared with the model performance of the novel model.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
According to private information law, the IPD generated and/or analyzed for this study will not be shared.

REFERENCES:
- [Background] Tay JK, Narasimhan B, Hastie T. Elastic Net Regularization Paths for All Generalized Linear Models. J Stat Softw. 2023;106:1. doi: 10.18637/jss.v106.i01. Epub 2023 Mar 23. PMID 37138589
- [Background] Park S, Park SH, Kim MS, Kwak J, Lee I, Kwon Y, Lee CM, Choi HS, Keum B, Yang KS, Park JM, Park S. Exploring objective factors to predict successful outcomes after laparoscopic Nissen fundoplication. Int J Surg. 2023 May 1;109(5):1239-1248. doi: 10.1097/JS9.0000000000000274. PMID 37026848
- [Background] Jung SW, Lee I, Lee I, Kim JW, Alromi A, Seo WJ, Park SH, Kwon Y, Jang YJ, Lee CM, Kim JH, Park JM, Park S. Bolus exposure as a novel predictor of postoperative symptom resolution after laparoscopic Nissen fundoplication: a two-institutional retrospective cohort study. Int J Surg. 2024 Dec 1;110(12):7919-7928. doi: 10.1097/JS9.0000000000002124. PMID 39453844
- [Background] Farrell TM, Richardson WS, Trus TL, Smith CD, Hunter JG. Response of atypical symptoms of gastro-oesophageal reflux to antireflux surgery. Br J Surg. 2001 Dec;88(12):1649-52. doi: 10.1046/j.0007-1323.2001.01949.x. PMID 11736981
- [Background] Yamasaki T, Fass R. Reflux Hypersensitivity: A New Functional Esophageal Disorder. J Neurogastroenterol Motil. 2017 Oct 30;23(4):495-503. doi: 10.5056/jnm17097. PMID 28992673
- [Background] Zhang D, Liu S, Li Z, Wang R. Global, regional and national burden of gastroesophageal reflux disease, 1990-2019: update from the GBD 2019 study. Ann Med. 2022 Dec;54(1):1372-1384. doi: 10.1080/07853890.2022.2074535. PMID 35579516